CLINICAL TRIAL: NCT02813421
Title: Professional Continuous Glucose Monitoring Before Starting Insulin Pump Therapy
Brief Title: Continue Glucose Monitoring Before Insulin Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jessica Ferris, MD, Clinical Fellow, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-15-00535
Record Dates: First submitted 2016-06-02; First posted 2016-06-27 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGM Informed (Experimental): CGM data was available for use when determining starting insulin pump doses.
  Interventions: Device: CGM Informed
- Control (No Intervention): CGM data will remain secure and not used. Starting insulin pump doses will be made by standard of care.

INTERVENTIONS:
Device: CGM Informed
  Other Names: iPro2 Professional Continuous Glucose Monitor
  Arms: CGM Informed

SUMMARY:
The purpose of the study is to learn more about blood glucose control when people with Type 1 Diabetes switch to an insulin pump. The investigators hope to learn whether using a continuous glucose monitor (CGM) helps to create personalized insulin doses that may lead to stable blood glucoses and less frequent insulin pump dose changes during the transition to an insulin pump.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled study. Participants will be asked to wear a Medtronic iPro2 continuous glucose monitor (CGM) 1-2 weeks prior to starting on insulin pump therapy. Depending on randomization groups, participants will either have CGM data used inform starting insulin pump doses (treatment group), or to standard of care for starting on insulin pump (control group). Participants will wear the CGM again during the first 5 days of pump start and at approximately 6 weeks after pump start, in order to collect blood glucose data. Each time the CGM is worn, blood glucoses must be checked 6-8 times daily, and a written log must be completed. Baseline medical information also will be collected at the start of participation. Participants will also be asked to complete a questionnaire at approximately 6 weeks after pump start. Participation in the study will be complete after a standard of care follow up visit approximately 3 months after pump start.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females aged 2-24 years
2. Clinical diagnosis of Type 1 diabetes mellitus
3. Duration of diabetes: At least 6 months

   - This will ensure some glycemic stability prior to study, and most children do not start on an insulin pump until about 6 months into their diagnosis.
4. Basal/bolus insulin regimen using long-acting and rapid-acting insulin

   - This will provide a uniform method of insulin therapy.
5. Willingness to perform at least 6-8 capillary blood glucose tests per day while wearing the iPro®2
6. Willingness to wear the iPro®2 for 5 days continuously per insertion
7. Participant agrees to comply with the study protocol requirements
8. Informed Consent, Assent, HIPAA Authorization, and California Experimental Subject Bill of Rights signed by the participant and/or parent guardian

Exclusion Criteria:

1. Comorbid conditions, including but not limited to cystic fibrosis, oncologic processes, other systemic diseases that may affect overall glycemic control
2. Glucocorticoid use within 2 weeks of study enrollment
3. Concurrent use of other medications that may affect glycemic control
4. Prior CGM use in the past 6 months
5. The participant has any skin abnormality (e.g. psoriasis, rash, staphylococcus infection) in the area of iPro®2 placement that has not been resolved at the time of enrollment and would inhibit the participant from wearing the iPro®2.
6. Non-English or non-Spanish speaking

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Ferris, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Informed: CGM data was available for use when determining starting insulin pump doses.
  CGM Informed
Period: Overall Study
Arm/Group | CGM Informed | Control
Started | 5 | 6
Completed | 3 | 3
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM Informed | Control | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (4.4) | 10.0 (3.0) | 10.6 (3.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 4 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: z-score] — BMI Z-score refers to standard deviation above the mean. Mean= 50%ile = z-score of 0, Negative value is SD below the mean, Positive value is SD above the mean.
  z-score | 1.36 (0.58) | 1.38 (0.6) | 1.37 (0.56)
Tanner Stage [Mean (Full Range); unit: Tanner Stage (1-5)] — Tanner stage represents pubertal stage. Tanner stage is a standardized measure to grade puberty on physical exam using a whole unit scale of 1 (pre-pubertal) through 5 (full pubertal). Insulin requires can differ depending on pubertal stage.
  Tanner Stage (1-5) | 3 [1 to 5] | 2 [1 to 4] | 3 [1 to 5]
Hemoglobin A1c (%) [Mean (Standard Deviation); unit: Percentage] | 7.6 (1.7) | 7.5 (0.94) | 7.55 (1.25)
Mean glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 173 (46) | 171 (38) | 172 (40)
Frequency of Blood Glucose Monitoring (times/day) [Mean (Standard Deviation); unit: Times/day] | 5.7 (2.6) | 6.7 (1.3) | 6.26 (1.99)
Age of Diagnosis (years) [Mean (Standard Deviation); unit: years] | 8 (4.2) | 8.1 (3.3) | 8.09 (3.56)
Duration of Diabetes (years) [Mean (Standard Deviation); unit: years] | 3.3 (4.9) | 1.8 (1.0) | 2.50 (3.27)
Daily Insulin dose (u/kg/day) [Mean (Standard Deviation); unit: units/kg/day] | 0.96 (0.55) | 0.72 (0.28) | 0.80 (0.42)
Daily Basal Insulin (%=percentage of total daily insulin dose that is used for basal insulin)) [Mean (Standard Deviation); unit: Percentage of total daily insulin] — Percentage of total daily insulin dose that is used for basal insulin
  Percentage of total daily insulin | 33.6 (10.2) | 40.2 (10.2) | 37.8 (11.7)
Episodes of DKA [Number; unit: Episodes] | 0 | 0 | 0
Population total number of episodes of significant hypoglycemia [Number; unit: Number of Episodes] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Time Within Target Blood Glucose (Range: 70-180 mg/dL)
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Percentage of time | 81.7 (13) | 68.0 (27)

2. Secondary Outcome: Percentage of Time Within Target Blood Glucose (Range: 70-180 mg/dL)
Time Frame: First 5 days of insulin pump therapy
Population: One control participant was lost to follow up after first 5 days of insulin pump therapy, therefore n=4 for this outcome, and not after.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 4
Percentage of time | 71 (8.2) | 57.5 (10.4)

3. Secondary Outcome: Mean Blood Glucose (mg/dL)
Description: Other measures of glycemic variability obtained by iPro2 download
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
mg/dL | 137 (6.6) | 193 (81)

4. Secondary Outcome: Percentage Time Hyperglycemic
Description: Data obtained by iPro2 download
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Percentage of time | 13.7 (9.7) | 31.7 (26)

5. Secondary Outcome: Total Daily Insulin Dose (Units)
Description: Will be obtained by insulin pump download.
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Units/kg/day | 0.88 (0.67) | 0.87 (0.53)

6. Secondary Outcome: Percentage Basal Insulin (%)
Description: Will be obtained by insulin pump download.
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Percentage of time | 34.5 (17) | 27.5 (4.8)

7. Secondary Outcome: Total Number of Insulin Dose Adjustments
Description: This data will be collected on standardized log sheets.
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Adjustments
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Adjustments | 18.7 (4.0) | 12.7 (11.2)

8. Secondary Outcome: Total Number of Phone Calls to Clinic Hotline
Description: This data will be collected on standardized log sheets.
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Phone calls
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Phone calls | 8.33 (3.51) | 5.67 (2.12)

9. Secondary Outcome: Number of Insulin Dose Adjustments Made Per Phone Call
Description: This data will be collected on standardized log sheets.
Time Frame: First 6 weeks of insulin pump therapy
Measure: Mean (Standard Deviation); unit: Changes/call
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Changes/call | 2.39 (0.55) | 1.96 (1.71)

10. Secondary Outcome: Episodes of DKA
Time Frame: First 6 weeks of insulin pump therapy
Measure: Number; unit: Episodes
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Episodes | 0 | 0

11. Secondary Outcome: Total Number of Episodes of Severe Hypoglycemia
Time Frame: First 6 weeks of insulin pump therapy
Measure: Number; unit: Number of Events
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Number of Events | 0 | 0

12. Secondary Outcome: Hemoglobin A1c (%)
Description: Difference in HbA1c from baseline to 3 months post-pump start
Time Frame: Baseline to 3 months post-pump start
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 3
Percentage of HbA1c | -0.27 (0.5) | 0.025 (0.67)

13. Secondary Outcome: Number of Participants With Satisfaction of Transition to Pump Therapy
Description: 6 question survey addressing patient/parent impressions of the process of transitioning to insulin pump therapy.
Time Frame: At 6 weeks after start of insulin pump therapy
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Informed | Control
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CGM Informed | Control
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02813421/Prot_SAP_000.pdf